CLINICAL TRIAL: NCT05922371
Title: ObsErvational Study of the Practical Cinical UTility of the NuQ.® H3.1 Nucleosome Levels in Adult Patients With Sepsis to Facilitate Early Diagnosis and Prognostication. (EPICETUS)
Acronym: EPICETUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Volition Diagnostics UK Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 324730
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sepsis: Adult patients admitted to critical care with a presumed diagnosis of sepsis.
  Interventions: Diagnostic Test: NuQ H3.1 Nucleosome Assay
- Cardiac surgery: Adult cardiac surgery patients that are free from infection undergoing their first cardiac surgery.
  Interventions: Diagnostic Test: NuQ H3.1 Nucleosome Assay

INTERVENTIONS:
Diagnostic Test: NuQ H3.1 Nucleosome Assay — Serial analysis on whole blood of nucleosome levels until resolution of sepsis or discharge.

SUMMARY:
This is a study to evaluate the diagnostic performance of the investigation NuQ. (R) H3.1 nucleosome assay as a diagnostic marker of sepsis in a population of patients admitted to critical care with signs suspicious of infection and consistent with the sepsis 3 definition. These patients will be compared to a group of adult surgical patients free from infection that are undergoing their first cardiac surgery.

DETAILED DESCRIPTION:
This is a single centre, prosepctive study to evaluate the diagnostic performance of the investigation NuQ. (R) H3.1 nucleosome assay as a diagnostic marker of sepsis in a population of patients admitted to critical care with signs suspicious of infection and consistent with the sepsis 3 definition. The H3.1 assay is a chemiluminescent sandwich immunoassay for the detection of nucleosomes circulating in human plasma. The test quantifies the level of circulating nucleosomes and in conjunction with other laboratory findings and clinical assessment aids in the early detection of sepsis with organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age to be included in the study.
* Patients must have been admitted to critical care emergently with signs and symptoms consistent with a possible diagnosis of sepsis: defined as one of these types of infections: respiratory system, renal and genito-urinary system, gastrointestinal and intra-abdominal system, central nervous system, musculoskeletal, sepsis or fever of unknown origin
* A 'comparator' arm will be included of patients aged over 18yrs of age undergoing planned elective coronary artery bypass graft surgery with anticipated post-operative care in critical care unit

Exclusion Criteria:

* Any subject not meeting the criteria above.
* Patients who are re-admitted to intensive care unit within the same hospital admission
* The exclusion criteria are designed to remove confounding effects from concomitant conditions that may render the interpretation of the NuQ.® H3.1 assay impossible. These circumstances are few, but exclusions will include patients with limitations of care, including 'Do not attempt resuscitation' orders.
* Patients with severe anaemia (as defined by a Hb<50g/dL) will be excluded.
* Subjects with any other severe concurrent disease that, in the judgment of the Principal Investigator, would make the subject inappropriate for entry into this study.
* Patients in the 'comparator' arm who are undergoing cardiac surgery will be excluded if they have an active infection and specifically patients with a suspected or confirmed diagnosis of infective endocarditis.
* Any patient undergoing cardiac surgery with a condition that might influence their immune response will be excluded. These include but are not limited to uncontrolled HIV, AIDS, uncontrolled systemic lupus erythematosus, rheumatoid arthritis or mixed connective tissue disorder, previous cancer and previous treatment with chemotherapy or the recipient of a solid organ or bone marrow transplant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited into two cohorts. The first cohort are patients who require critical care admission emergently from either A&E or other hospital ward with a presumed diagnosis of sepsis. The second group consists of patients who have a planned elective cardiac surgery (Coronary Artery By-Pass Graft surgery) and require critical care admission post operatively as part of the planned surgery. These patients have been selected to describe how the level of NuQ.® H3.1 alters over time after the sterile insult of cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the levels of H3.1 nucleosomes in critically ill patients diagnosed with sepsis. | 14 days
  To investigate the levels of H3.1 nucleosomes in critically ill patients diagnosed with sepsis or septic shock (as defined by Sepsis-3 criteria at time of presentation), specifically to monitor how these levels change over time in relation to disease progression, clinical data and other routinely collected biomarkers such as CRP and procalcitonin.

SECONDARY OUTCOMES:
To investigate the potential utility of levels of NETs/Cf DNA (as measured by the H3.1 nucleosome assay) as a companion diagnostic test of septic shock, disease monitoring, severity and prognosis. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided